CLINICAL TRIAL: NCT01266551
Title: The Car Safety Seat; Cause of Increased Gastroesophageal Reflux Disease in Infants?
Brief Title: Car Safety Seat and Gastroesophageal Reflux Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intended number of patients reached
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 3204
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2008-10

CONDITIONS: Gastroesophageal Reflux Disease and Position
Keywords: Antireflux procedure; Gastroesophageal reflux; Infant sleep position; pH monitoring
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counseling (No Intervention): The positions in the car safety seat and in supine 15 degrees anti-Trendelenburg are compared on the basis of a 20 hour pH monitoring. In one group the infants were first continuously positioned at 45 degrees elevation in a car safety seat (car safety seat type Maxi cosi Citi for infants from 0-13kg). During the next period the infants were kept in a supine 15 degrees anti-Trendelenburg position (hospital infant bed), and vice versa for the other group.
  Interventions: Device: car safety seat

INTERVENTIONS:
Device: car safety seat — The positions in the car safety seat and in supine 15 degrees anti-Trendelenburg are compared on the basis of a 20 hour pH monitoring.In one group the infants were first continuously positioned at 45 degrees elevation in a car safety seat (car safety seat type Maxi cosi Citi for infants from 0-13kg). During the next period the infants were kept in a supine 15 degrees anti-Trendelenburg position (hospital infant bed), and vice versa for the other group.

SUMMARY:
What's known? Prone position is no longer a treatment option for GERD because of the association with SIDS. Originally, positioning in an infant seat was recommended for infants with GERD. However, Orenstein proved this position has a detrimental effect on GER, compared to prone positioning.

What's new? Positioning in an infant seat caused no increase in GER, compared with the supine 15 degrees anti-Trendelenburg position. Except for the number of long reflux episodes, which was significantly higher in the car safety seat. Larger trials are needed for decisive conclusions.

DETAILED DESCRIPTION:
OBJECTIVE - Over the past few decades, an increase in gastroesophageal reflux disease (GERD) has been seen in infants. This increase may be due to a continuous growth in the use of car safety seats. The objective of this study was to evaluate this hypothesis by comparing positioning in a car safety seat with the supine 15 degrees anti-Trendelenburg position.

PATIENTS AND METHODS - From October 2008 till August 2010 a crossover, randomized, controlled trial was performed on 31 infants, aged two weeks to six months old, who were suspected to have GERD. Twenty hour continuous esophageal pH monitoring was used to compare both positions.

RESULTS - The results of this trial demonstrated no differences between positioning in a car safety seat and in supine 15 degrees anti-Trendelenburg position for the reflux index, the duration of the longest reflux episode and number of reflux episodes (PRI = NS; PLRE = NS respectively PNRE = NS). Only the difference between the number of reflux episodes lasting longer than five minutes was significant (PNRE5 = 0,05).

CONCLUSIONS - The results of this study suggest that an increase in GERD is not caused by a growing use of car safety seats in infants. As the sample size was limited, larger trials are needed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: healthy term-born infants between two weeks and six months old suspected to have GERD, in general good health. The infants did not need to meet the criteria for GERD to be eligible.

Exclusion Criteria:

* Exclusion criteria were infants with psychomotor retardation, acute illness or contra-indication for pH monitoring.

Ages: 2 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2008-10 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, Belgium